CLINICAL TRIAL: NCT04145752
Title: Acute Pain in Hip Fracture Patients: Pain Management in the Emergency Department, a Mixed Method Study¨. Nurse Led Ultrasound Guided Femoral Nerve Block in the Emergency Department
Brief Title: Nurse Led Ultrasound Guided Femoral Nerve Block in the Emergency Department
Acronym: URGENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Espen Lindholm (Other)
Collaborators: University College of Southeast Norway (Other)
Responsible Party: Sponsor-Investigator, Espen Lindholm, Senior consultant, Sykehuset i Vestfold HF
Organization: Sykehuset i Vestfold HF (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: URGENT 2019
Record Dates: First submitted 2019-10-25; First posted 2019-10-31 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Hip Fractures; Anesthesia; Femoral Neck Fractures
Keywords: femoral nerve block; Ultrasound guided; Nurse-led
MeSH Terms: conditions — Hip Fractures; Femoral Neck Fractures

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, controlled, open label trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurse-led femoral nerve block (Experimental): Trained nurses in ED provide ultrasound guided single-shot femoral nerve block shortly after (at arrival emergency department) the patient is diagnosed with a hip fracture.
  Drug: Ropivacaine 3 mg/kg, single-shot
  Interventions: Procedure: Nurse-led femoral nerve block
- Standard of care (Active Comparator): Nurses do not provide ultrasound guided single-shot FNB and the patient follows the standard of care course.
  Interventions: Procedure: Nurse-led femoral nerve block

INTERVENTIONS:
Procedure: Nurse-led femoral nerve block — The nurse perform a femoral nerve block in the emergency department in patients diagnosed with a hip fracture (x-ray)

SUMMARY:
The aim of this study is to investigate the effects of task shifting from anesthesiologists to special trained nurses performing femoral nerve block (FNB) in patients with hip fracture in the emergency department (ED) at Vestfold Hospital Trust (VHT). A sample of nurses (n= 6) will perform ultrasound guided FNB in hip fracture patients (n=25) admitted to the ED at VHT. This cohort will be compared to another cohort of hip fracture patients (n=25). This cohort will follow standard of care where the femoral nerve block is often performed by anesthesiologists. The study is a prospective, controlled randomized trial.

DETAILED DESCRIPTION:
The ageing population admitted to the ED in developed countries is steadily increasing. Hip fractures are common among the elderly population, and related to increased mortality. Patient satisfaction with ED's has been an international challenge over several years. Acute pain is one of the most common reasons for patients coming admitted to the ED. However, undertreatment of pain is common, particularly in patients with hip fractures.

Pain control can be difficult, and often requires intensive nursing and physician care, as elderly patients may manifest cardiovascular and respiratory complications from opioid administration. Optimizing acute pain management in patients with orthopedic trauma is important and can translate into significant positive physiologic and financial outcomes.

At Vestfold Hospital Trust, pain relief of the hip fracture patient in ED has traditionally most often consisted of paracetamol and opiates. Additionally, the patients are offered FNB by the anesthesiologist, but concurrent conflicts and other organizational circumstances has have led to delayed block or no block for all or some patients. This often necessitate a continuation of pain relief in form of intravenous opioids, with increased risk of opioid side effects such as respiratory depression, delirium, constipation, urinary retention, nausea and vomiting and subsequently increased morbidity and increased costs for the hospital and the community.

The investigators believe that shifting this task to nurses working in the ED can secure patient with hip fractures sufficiently and timely pain relief. By giving trained nurses this new task of performing FNB the investigators can study how expert nurses qualifications' are utilized to strengthen the quality of the ED. This study aims to implement and evaluate the introduction of specially trained nurses performing ultrasound guided FNB in patients with hip fractures in the ED. This implementation may be beneficial to patients in terms of prompt analgesia, reduced opioid consumption, thereby reducing opioid adverse events, and it might influence risk of complications and length of stay. The aim of this study is to evaluate cumulative Numeric Rating Scale (NRS) score during rest and during passive movement (30 degree flexion in the hip) in patients with hip fracture during stay in the ED at 120 minutes after admission, thereby comparing nurse-led FNB versus standard of care.

The study has a randomized controlled trial design. Patients are randomized (1:1) into two groups:

1. Trained nurses in ED provide ultrasound guided single-shot FNB shortly after (at arrival ED) the patient is diagnosed with a hip fracture.
2. Nurses do not provide ultrasound guided single-shot FNB and the patient follows the FAST-TRACK-HIP FRACTURE course local guideline at our hospital.

Hypothesis: A single shot FNB performed by nurses in the ED compared to todays practice will result in lower cumulative NRS score first 120 minutes after admission to ED than current practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients arriving at the emergency department diagnosed with a hip fracture (X-ray confirmed)
* American Society of Anesthesiologists classification (ASA) 1-4
* Written informed consent by patient

Exclusion Criteria:

* Patients with dementia
* Known allergies to local anesthetic used in femoral nerve block.
* The patient is anticoagulated or uses platelet inhibitors. Acetylsalicylic acid and dipyridamole is allowed. If a recent (last 2 hours) International normalized ratio (INR) is below <1.5 the patient can be included.
* Pregnant
* Age <18 years
* Severe head injury which leads to significant loss of consciousness (Glascow coma score (GCS) <12)
* >10 mg or more morphine administrated pre-hospital
* Skin lesions/infection at block site
* Patients admitted with other suspected or verified fractures, except small fractures in hands and foots.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Cumulative dynamic pain score - Numerical Rating Scale (NRS) - during passive movement at 120 minutes after start of procedure | 120 minutes
  Cumulative dynamic pain score - Numerical Rating Scale (NRS) - during passive movement (30 degree flexion in the fractured hip) in patients with hip fracture during stay in the ED at 120 minutes after admission, measured by five time Points; At the end of procedure, 30 min.-, 60 min.-, 90 min.- and 120 min after start of procedure. NRS score: 0 is no pain and 10 is the worst pain.

SECONDARY OUTCOMES:
Number of total morphine equivalents - 24h | 24 hours
  Number of total morphine equivalents, mg (iv/po) administered during first 24 hours from admission at the emergency department
Number of total morphine equivalents - Hospital stay | approx. 6 days
  Number of total morphine equivalents, mg (iv/po) administered during total hospital stay.
Cumulative rest pain score -Numerical Rating Scale (NRS) - at 120 minutes after start of procedure | 120 minutes
  Cumulative rest pain score NRS - Numerical Rating Scale (NRS) - in patients with hip fracture during stay in the emergency department at 120 minutes after admission, measured by five time Points; At the end of procedure, 30 min.-, 60 min.-, 90 min.- and 120 min after start of procedure. NRS score: 0 is no pain and 10 is the worst pain.

OTHER OUTCOMES:
Incidence of delirium during hospital stay. | Approx. 6 days
  Incidence of delirium, measured by Assessment test for delirium & cognitive impairment - 4AT, will be performed daily during hospital stay, number of patients
RASS-score - Richmond Agitation and Sedation Scale | Daily - approx. 6 days
  Measure consciousness assessed by RASS-score - Richmond Agitation and Sedation Scale - (at admittance to the emergency department and daily). Total score. RAAS is a10-point scale, with four levels of anxiety or agitation (+1 to +4), one level to denote a calm and alert state (0), and 5 levels of sedation (-1 to -5) culminating in unarousable (-5).
Number of (mg) administered of antiemetics during hospital stay | approx. 6 days
  Number of (mg) administered of antiemetics ( ondansetron, dexagalen, metoclopramide) during first 24 hours and during hospital stay.
Time (minutes) to perform an ultrasound guided femoral nerve block performed | approx 30 minutes
  Time (minutes) used to perform an ultrasound guided femoral nerve block performed by nurses.
Time from arrival at the emergency department to femoral nerve block is performed | Approx 1 hour
  Time (min.) from arrival at emergency department (from Radiological Department) to femoral nerve block is performed.
Time from admission to surgery starts | approx. 48 hours
  Time from admission to surgery starts, minutes
Length of total hospital stay | Approx. 6 days
  Length of total hospital stay, days
Mortality during hospitalization | Approx. 6 days
  Mortality during hospitalization, Yes or no
Mortality 30 days | 30 days
  Mortality at postoperative day 30, Yes or no
Hospital acquired pneumonia | Approx 6 days
  Hospital acquired pneumonia during hospital stay, Yes or no
Acute myocardial infarction | Approx 6 days
  Acute myocardial infarction during hospital stay, Yes or no
Acute renal failure | Approx 6 days
  Acute renal failure during hospital stay, Yes or no
Respiratory failure | Approx 6 days
  Respiratory failure during hospital stay, Yes or no
Intravasal injection | 24 hours
  Intravasal injection - visually + circulatory and neurological symptoms, Yes or no
Hematoma | 24 hours
  Hematoma - defined as a new tumor > 2 centimeter in the groin / injection site measured by ultrasound, Yes or no
Neurologic systemic outcomes / symptoms / paresthesia | Approx 6 days
  Neurologic systemic outcomes / symptoms / paresthesia that have occurred after admission and which persist until discharge, numbers

CONTACTS AND LOCATIONS:
Overall Officials: Elin Saga, nurse, Principal Investigator — The Hospital of Vestfold
Locations (1):
- Sykehuset i Vestfold HF, Tønsberg, Norway

IPD SHARING:
Plan to Share IPD: No
No plan at this moment

REFERENCES:
- [Derived] Saga E, Falk RS, Bing-Jonsson PC, Skovdahl KI, Lindholm E. Nurse-led ultrasound-guided femoral nerve block: A randomised controlled trial of two different patient flow systems in an emergency department. Int J Orthop Trauma Nurs. 2024 Feb;52:101074. doi: 10.1016/j.ijotn.2023.101074. Epub 2023 Dec 4. PMID 38070309
- [Derived] Guay J, Kopp S. Peripheral nerve blocks for hip fractures in adults. Cochrane Database Syst Rev. 2020 Nov 25;11(11):CD001159. doi: 10.1002/14651858.CD001159.pub3. PMID 33238043